CLINICAL TRIAL: NCT06843889
Title: A Phase II Study of Toripalimab Combined With Sequential Neoadjuvant Chemoradiotherapy in Patients With Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2025-054
Record Dates: First submitted 2025-02-18; First posted 2025-02-25 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma
Keywords: Esophageal cancer; Immunotherapy; Neoadjuvant radiotherapy; Neoadjuvant chemotherapy; Efficacy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy combined with sequential neoadjuvant radiotherapy group (Experimental)
  Interventions: Drug: Toripalimab (240mg day1, Q3W*3cycle)

INTERVENTIONS:
Drug: Toripalimab (240mg day1, Q3W*3cycle) — Phase 1: Toripalimab (240mg day1, Q3W*2cycle) + investigator's choice of clinical conventional chemotherapy; Phase 2: Toripalimab (240mg day1, Q3W*1cycle) + radiotherapy (intensity modulated radiotherapy, 40Gy/20F, 2Gy/F); Surgery was performed 4-6 weeks after completion, and subsequent treatment options were considered after surgery according to MDT discussion.

SUMMARY:
This was a single-center, open phase II clinical study. 34 patients with resectable local middle and advanced esophageal squamous cell carcinoma were treated with anti-PD-1 antibody combined with sequential chemoratherapy regimen: Phase I:Toripalimab (240mg day1, Q3W*2cycle) + clinical routine chemotherapy regimen selected by the investigator; The second stage: Toripalimab (240mg day1, Q3W*1cycle) + radiotherapy (intensity modulated radiotherapy, 40Gy/20F, 2Gy/F); Surgery was performed 4-6 weeks after completion, and subsequent treatment options were considered after surgery according to MDT discussion. According to the postoperative pathological results, the pathological complete response (pCR) and major response (MPR) were evaluated. The disease-free survival (DFS), overall survival (OS), 1 or 2 years survival rate and adverse reactions were recorded.

ELIGIBILITY:
Inclusion Criteria:

* 1: age 18-75 years old, both sexes; 2: esophageal squamous cell carcinoma confirmed by histopathology; 3: T2-4a, N0-3, M0 (AJCC 8th edition) thoracic esophageal cancer patients, resectable by surgical evaluation; 4: initial treatment patients without anti-tumor therapy; 5: expected survival time ≥6 months; 6: ECOG ≤1; 7: There was no history of esophageal perforation, active esophageal bleeding, and no obvious invasion of trachea or thoracic large vessels.

  8: The function of vital organs meets the following requirements: white blood cell ≥4.0×109/l, neutrophil ≥1.5×109/l, platelet ≥100.0×109/l, hemoglobin ≥90g/l; Serum albumin ≥2.8g/Dl; Total bilirubin ≤1.5 × ULN, ALT/AST/ AKP≤2.5 × ULN; Serum creatinine ≤1.5 × ULN or creatinine clearance > 60 mL/min; There were no severe organic diseases.

  9: FEV1 ≥ 0.8L; 10: Patients were informed about the trial details and signed informed consent.

Exclusion Criteria:

* 1: known to be allergic to recombinant humanized anti-PD-1 monoclonal antibody drugs or their components; 2: currently participating in and receiving other study treatment; 3: previous systemic therapy for esophageal cancer, including systemic chemotherapy, targeted therapy, immunotherapy, etc.

  4: patients with active pulmonary tuberculosis (TB) who were receiving anti-TB treatment or received anti-TB treatment within 1 year before screening; 5: uncontrolled or symptomatic hypercalcemia (>1.5mmol/L calcium ion or calcium >12mg/dL or corrected serum calcium >ULN); 6: clinically uncontrolled active infection, including but not limited to acute pneumonia; 7: uncontrolled major seizures or superior vena cava syndrome; 8: previous or current concomitant other malignant tumors (except non-melanoma basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the breast/cervix, superficial bladder, etc., which were treated radically and had no evidence of disease recurrence) 9: Patients with a history of interstitial pneumonia, idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, evidence of active pneumonia detected by chest CT scan or other moderate to severe lung diseases that seriously affect lung function; 10: known human immunodeficiency virus (HIV) infection (known HIV antibody positive); 11: severe cardiovascular disease, such as New York Heart Association (NYHA) class 2 or higher heart failure, unstable angina, unstable arrhythmia, myocardial infarction or cerebrovascular accident within 6 months before enrollment; 12: received systemic immunosuppressive drugs (i.e., corticosteroids or immunosuppressive drugs) for any active autoimmune disease within 2 years before study entry; 13: received live viral vaccine within 4 weeks before study entry; 14: patients with prior allogeneic stem cell or solid organ transplantation; 15: pregnant or lactating women or women with the possibility of pregnancy before the first medication positive pregnancy test, patients with fertility but unwilling to accept contraceptive measures or their sexual partners unwilling to accept contraceptive measures; 16: any other disease or condition of clinical significance that the investigator believes could affect adherence to the protocol (e.g., history of psychosis or substance abuse), preclude benefit from the study, or prevent informed consent (e.g., drug use and substance abuse), or preclude participation in the study (including but not limited to: Abnormal laboratory results, clinical active diverticulitis, intra-abdominal abscess, intestinal obstruction, and peritoneal carcinomatosis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response Rate (pCR) | Perioperative
  The absence of residual viable tumor cells in both the primary esophageal tumor and regional lymph nodes after completion of neoadjuvant chemoradiotherapy and surgery, indicating a complete pathological response.

SECONDARY OUTCOMES:
Major Pathological Response Rate (MPR) | Perioperative
  A significant reduction in tumor burden, defined as less than 10% residual viable tumor in the surgical specimen following neoadjuvant chemoradiotherapy, reflecting a near-complete response.
Disease-Free Survival (DFS) | From the date of surgery (or completion of treatment) to the date of the first documented disease recurrence, metastasis, or death from any cause, whichever occurred first,assessed up to 100 months.
  The duration from the date of surgery to the first occurrence of disease recurrence, metastasis, or death from any cause, measuring the effectiveness of the treatment in preventing disease progression.
Overall Survival (OS) | From the date of treatment initiation (or diagnosis) to the date of death from any cause,assessed up to 120 months..
  The length of time from the start of neoadjuvant treatment until death from any cause, evaluating the long-term survival benefit of the combined therapy.
Adverse Events (AEs) | Monitored throughout the treatment period and during follow-up, an average of 2 years.
  Any unfavorable or unintended medical occurrences, including clinical signs, symptoms, or laboratory abnormalities, observed in patients receiving toripalimab combined with neoadjuvant chemoradiotherapy, regardless of causality.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Baiyun District, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Sharma P, Allison JP. The future of immune checkpoint therapy. Science. 2015 Apr 3;348(6230):56-61. doi: 10.1126/science.aaa8172. PMID 25838373
- [Background] Ford HE, Marshall A, Bridgewater JA, Janowitz T, Coxon FY, Wadsley J, Mansoor W, Fyfe D, Madhusudan S, Middleton GW, Swinson D, Falk S, Chau I, Cunningham D, Kareclas P, Cook N, Blazeby JM, Dunn JA; COUGAR-02 Investigators. Docetaxel versus active symptom control for refractory oesophagogastric adenocarcinoma (COUGAR-02): an open-label, phase 3 randomised controlled trial. Lancet Oncol. 2014 Jan;15(1):78-86. doi: 10.1016/S1470-2045(13)70549-7. Epub 2013 Dec 10. PMID 24332238
- [Background] Ross P, Nicolson M, Cunningham D, Valle J, Seymour M, Harper P, Price T, Anderson H, Iveson T, Hickish T, Lofts F, Norman A. Prospective randomized trial comparing mitomycin, cisplatin, and protracted venous-infusion fluorouracil (PVI 5-FU) With epirubicin, cisplatin, and PVI 5-FU in advanced esophagogastric cancer. J Clin Oncol. 2002 Apr 15;20(8):1996-2004. doi: 10.1200/JCO.2002.08.105. PMID 11956258
- [Background] Shah MA, Janjigian YY, Stoller R, Shibata S, Kemeny M, Krishnamurthi S, Su YB, Ocean A, Capanu M, Mehrotra B, Ritch P, Henderson C, Kelsen DP. Randomized Multicenter Phase II Study of Modified Docetaxel, Cisplatin, and Fluorouracil (DCF) Versus DCF Plus Growth Factor Support in Patients With Metastatic Gastric Adenocarcinoma: A Study of the US Gastric Cancer Consortium. J Clin Oncol. 2015 Nov 20;33(33):3874-9. doi: 10.1200/JCO.2015.60.7465. PMID 26438119
- [Background] Day FL, Leong T, Ngan S, Thomas R, Jefford M, Zalcberg JR, Rischin D, McKendick J, Milner AD, Di Iulio J, Matera A, Michael M. Phase I trial of docetaxel, cisplatin and concurrent radical radiotherapy in locally advanced oesophageal cancer. Br J Cancer. 2011 Jan 18;104(2):265-71. doi: 10.1038/sj.bjc.6606051. Epub 2010 Dec 14. PMID 21157450
- [Background] Li QQ, Liu MZ, Hu YH, Liu H, He ZY, Lin HX. Definitive concomitant chemoradiotherapy with docetaxel and cisplatin in squamous esophageal carcinoma. Dis Esophagus. 2010 Apr;23(3):253-9. doi: 10.1111/j.1442-2050.2009.01003.x. Epub 2009 Aug 28. PMID 19732130
- [Background] Urba SG, Orringer MB, Ianettonni M, Hayman JA, Satoru H. Concurrent cisplatin, paclitaxel, and radiotherapy as preoperative treatment for patients with locoregional esophageal carcinoma. Cancer. 2003 Nov 15;98(10):2177-83. doi: 10.1002/cncr.11759. PMID 14601087
- [Background] Kang YK, Kang WK, Shin DB, Chen J, Xiong J, Wang J, Lichinitser M, Guan Z, Khasanov R, Zheng L, Philco-Salas M, Suarez T, Santamaria J, Forster G, McCloud PI. Capecitabine/cisplatin versus 5-fluorouracil/cisplatin as first-line therapy in patients with advanced gastric cancer: a randomised phase III noninferiority trial. Ann Oncol. 2009 Apr;20(4):666-73. doi: 10.1093/annonc/mdn717. Epub 2009 Jan 19. PMID 19153121
- [Background] Bouche O, Raoul JL, Bonnetain F, Giovannini M, Etienne PL, Lledo G, Arsene D, Paitel JF, Guerin-Meyer V, Mitry E, Buecher B, Kaminsky MC, Seitz JF, Rougier P, Bedenne L, Milan C; Federation Francophone de Cancerologie Digestive Group. Randomized multicenter phase II trial of a biweekly regimen of fluorouracil and leucovorin (LV5FU2), LV5FU2 plus cisplatin, or LV5FU2 plus irinotecan in patients with previously untreated metastatic gastric cancer: a Federation Francophone de Cancerologie Digestive Group Study--FFCD 9803. J Clin Oncol. 2004 Nov 1;22(21):4319-28. doi: 10.1200/JCO.2004.01.140. PMID 15514373
- [Background] Al-Batran SE, Hartmann JT, Probst S, Schmalenberg H, Hollerbach S, Hofheinz R, Rethwisch V, Seipelt G, Homann N, Wilhelm G, Schuch G, Stoehlmacher J, Derigs HG, Hegewisch-Becker S, Grossmann J, Pauligk C, Atmaca A, Bokemeyer C, Knuth A, Jager E; Arbeitsgemeinschaft Internistische Onkologie. Phase III trial in metastatic gastroesophageal adenocarcinoma with fluorouracil, leucovorin plus either oxaliplatin or cisplatin: a study of the Arbeitsgemeinschaft Internistische Onkologie. J Clin Oncol. 2008 Mar 20;26(9):1435-42. doi: 10.1200/JCO.2007.13.9378. PMID 18349393
- [Background] Lorenzen S, Schuster T, Porschen R, Al-Batran SE, Hofheinz R, Thuss-Patience P, Moehler M, Grabowski P, Arnold D, Greten T, Muller L, Rothling N, Peschel C, Langer R, Lordick F. Cetuximab plus cisplatin-5-fluorouracil versus cisplatin-5-fluorouracil alone in first-line metastatic squamous cell carcinoma of the esophagus: a randomized phase II study of the Arbeitsgemeinschaft Internistische Onkologie. Ann Oncol. 2009 Oct;20(10):1667-73. doi: 10.1093/annonc/mdp069. Epub 2009 Jun 23. PMID 19549707